CLINICAL TRIAL: NCT00773747
Title: An International, Multicenter, Randomized, Double-Blind Study of Vorinostat (MK-0683) or Placebo in Combination With Bortezomib in Patients With Multiple Myeloma
Brief Title: Study of Vorinostat (MK-0683) or Placebo, in Combination With Bortezomib in Participants With Multiple Myeloma (MK-0683-088 AMN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0683-088; MK-0683-088 (Other: Merck Protocol Number); 2008-003752-30 (EudraCT Number)
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma
Keywords: Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Hemostatic Disorders; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases; Vorinostat; Bortezomib; Anti-Inflammatory Agents, Non-Steroidal; Analgesics, Non-Narcotic; Analgesics; Sensory System Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Pharmacologic Actions; Anti-Inflammatory Agents; Therapeutic Uses; Antirheumatic Agents; Antineoplastic Agents; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Anticarcinogenic Agents
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Hemostatic Disorders; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases | interventions — Vorinostat; Bortezomib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vorinostat + Bortezomib (Experimental): Participants will receive vorinostat four 100 mg capsules (400 mg total) orally 0-30 minutes after a meal on Days 1-14 of a 21-day treatment cycle and bortezomib 1.3 mg/m^2 by intravenous injection on Days 1, 4, 8, and 11 of a 21-day treatment cycle.
  Interventions: Drug: Vorinostat; Drug: bortezomib
- Placebo + Bortezomib (Placebo Comparator): Participants will receive four placebo capsules orally 0-30 minutes after a meal on Days 1-14 of a 21-day treatment cycle and bortezomib 1.3 mg/m^2 by intravenous injection on Days 1, 4, 8, and 11 of a 21-day treatment cycle.
  Interventions: Drug: bortezomib; Drug: placebo to vorinostat

INTERVENTIONS:
Drug: Vorinostat — Four 100 mg capsules vorinostat taken orally, once daily, on Days 1 through 14 of each 21-day treatment cycle.
  Other Names: Zolinza
  Arms: Vorinostat + Bortezomib
Drug: bortezomib — 1.3 mg/m2 of bortezomib by IV push, on Days 1, 4, 8, and 11 of each 21-day treatment cycle.
  Other Names: Velcade
Drug: placebo to vorinostat — Four placebo capsules taken orally, once daily, on Days 1 through 14 of each 21-day treatment cycle.
  Arms: Placebo + Bortezomib

SUMMARY:
Study of the efficacy and safety of bortezomib administered in combination with vorinostat in patients with relapsed or refractory multiple myeloma. Histone deacetylases (HDAC) facilitate gene transcription by modulating the uncoiling of chromatin. HDAC function is dysregulated in hematologic and solid malignancies, and this dysregulation may result in over-expression of oncogenes. Thus, inhibition of HDACs may result in anti-cancer effects. HDAC inhibitors, like vorinostat, represent a new class of antitumor agents that have the ability to induce antiproliferative effects including cyto-differentiation, cell cycle growth arrest or apoptosis in various cancer cell lines. Several studies have investigated the in vitro antimyeloma activity of vorinostat in combination with bortezomib and have demonstrated that vorinostat may act synergistically with bortezomib to modulate tumor cell growth. Mitsiades et al have shown that vorinostat enhances the sensitivity of bortezomib. Pei et al found that exposure of human multiple myeloma cell lines & patient-derived multiple myeloma cells to bortezomib and vorinostat resulted in synergistic interactions as a result of: (1) Interruption of NF-kB & related signaling pathways (JNK, XIAP, Mcl-1, etc.) (2) Inhibition of Hsp90 (3)Induction of ER stress signal and (4) acetylation of Dynein/disruption of aggresome function/formation, salvage for ubiquitinated proteins. In addition a marked increase in mitochondrial injury, caspase activation, and apoptosis was also observed. Bortezomib is indicated for the treatment of patients with multiple myeloma. Two Phase I dose-ranging studies of a regimen combining vorinostat and bortezomib among patients with relapsed as well asend-stage, refractory multiple myeloma have been conducted. These studies enrolled a total of 57 patients. In these studies, administration of vorinostat with standard doses of bortezomib resulted in responses in 20/45 (44%) evaluable patients (Weber et al 2007, Badros et al 2007). The purpose of the present study is to definitively evaluate the clinical activity of vorinostat in combination with bortezomib inpatients with multiple myeloma.

ELIGIBILITY:
Inclusion criteria

* Participant has an established diagnosis of multiple myeloma based on the myeloma diagnostic criteria.
* Participant has received at least 1 but not more than 3 prior anti-myeloma regimens and has progressive disease after the most recent treatment regimen.
* Participant must have adequate organ function.

Exclusion criteria:

* Participant has had a prior allogeneic bone marrow transplant or plans to undergo any type of bone marrow transplantation within 4 weeks of the initiation of study therapy.
* Participant has known hypersensitivity to any components of bortezomib or vorinostat.
* Participant has active Hepatitis B or C, plasma cell leukemia, or is human immunodeficiency virus (HIV) positive.
* Participant has had prior treatment with vorinostat or histone deacetylase (HDAC) inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2011-09-08 (Actual); Study Completion 2015-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Dimopoulos M, Siegel DS, Lonial S, Qi J, Hajek R, Facon T, Rosinol L, Williams C, Blacklock H, Goldschmidt H, Hungria V, Spencer A, Palumbo A, Graef T, Eid JE, Houp J, Sun L, Vuocolo S, Anderson KC. Vorinostat or placebo in combination with bortezomib in patients with multiple myeloma (VANTAGE 088): a multicentre, randomised, double-blind study. Lancet Oncol. 2013 Oct;14(11):1129-1140. doi: 10.1016/S1470-2045(13)70398-X. Epub 2013 Sep 19. PMID 24055414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants with an established diagnosis of multiple myeloma based on standard criteria that have received at least 1 but not more than 3 prior anti-myeloma regimens and have demonstrated progressive disease after the most recent treatment regimen. Additional inclusion and exclusion criteria applied.
Pre-assignment Details: 637 participants were randomized to treatment and 635 participants received at least 1 dose of MK-0683 or placebo: 315 participants were treated with vorinostat + bortezomib and 320 participants were treated with placebo + bortezomib.
Groups:
- Vorinostat + Bortezomib: Participants will receive vorinostat four 100 mg capsules (400 mg total) orally 0-30 minutes after a meal on Days 1 through 14 of a 21-day treatment cycle and bortezomib 1.3 mg/m^2 by intravenous injection on Days 1, 4, 8, and 11 of a 21-day treatment cycle.
- Placebo + Bortezomib: Participants will receive four placebo capsules orally 0-30 minutes after a meal on Days 1 through 14 of a 21-day treatment cycle and bortezomib 1.3 mg/m^2 by intravenous injection on Days 1, 4, 8, and 11 of a 21-day treatment cycle.
Period: Overall Study
Arm/Group | Vorinostat + Bortezomib | Placebo + Bortezomib
Started | 317 | 320
Treated | 315 | 320
Completed | 20 | 24
Not Completed | 297 | 296
Not completed — Lack of Efficacy | 112 | 144
Not completed — Physician Decision | 26 | 18
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 89 | 61
Not completed — Adverse Event | 61 | 62
Not completed — Death | 5 | 8
Not completed — Not Treated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorinostat + Bortezomib | Placebo + Bortezomib | Total
Number analyzed (Participants) | 317 | 320 | 637
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (10.0) | 62.7 (10.0) | 61.8 (10.0)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 200 | 181 | 381
  From 65-84 years | 116 | 137 | 253
  85 years and over | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 134 | 260
  Male | 191 | 186 | 377
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 23 | 55
  Not Hispanic or Latino | 285 | 297 | 582
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival was measured from the start of the treatment to the time when the criteria for progression was met or death due to any cause (whichever is first recorded). Response to study therapy was assessed using European Blood and Marrow Transplantation Group (EBMT) Criteria. A stratified Cox proportional hazards model was used with Efron's likelihood approximation to account for ties in event times.
Time Frame: From randomization to event of disease progression or death assessed up to 32 months (final study analysis)
Population: The analysis population includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vorinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 317 | 320
Months | 7.63 (6.87) [6.87 to 8.40] | 6.83 (5.67) [5.67 to 7.73]
Statistical Analysis 1: Comparison: Vorinostat + Bortezomib vs Placebo + Bortezomib; Cox model stratified by myeloma stage at enrollment, history of a bone marrow transplant, and number of prior treatment regimens, with a single treatment covariate; Test type: Superiority; p = 0.0100, Regression, Cox; Cox Proportional Hazard = 0.774, 95% CI 2-sided [0.636 to 0.941]

2. Secondary Outcome: Number of Participants With Grade 3-5 Clinical or Laboratory Adverse Events (AEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. Grades come from the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Per protocol, clinical and laboratory AEs are presented as a combined total for each grade.
Time Frame: Up to 722 days
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 315 | 320
Participants
  Grade 3 | 272 | 240
  Grade 4 | 108 | 85
  Grade 5 | 11 | 17

3. Secondary Outcome: Overall Survival
Description: Overall survival was measured from the start of the treatment to death due to any cause. Overall Survival is represented as the number of deaths per 100-person- months and was computed by dividing the number of participants with an event of death that occurred during the study follow-up period by the total duration of follow-up (in 100 months) for all the participants in each cohort since participants had different lengths of follow-up.
Time Frame: From randomization up to 32 months (final study analysis)
Population: The analysis population includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: Events/100-person Months
Arm/Group | Vorinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 317 | 320
Events/100-person Months | 1.7 (1.56) [1.56 to 1.84] | 1.9 (1.75) [1.75 to 2.05]
Statistical Analysis 1: Comparison: Vorinostat + Bortezomib vs Placebo + Bortezomib; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3496, Regression, Cox; Cox Proportional Hazard = 0.858, 95% CI 2-sided [0.622 to 1.184]

4. Secondary Outcome: Time to Progression
Description: Time to progression was measured from the start of the treatment to the time when the criteria for progression was met or death due to myeloma (whichever is first recorded). Response to study therapy was assessed using European Blood and Marrow Transplantation Group (EBMT) Criteria. A stratified Cox proportional hazards model was used with Efron's likelihood approximation to account for ties in event times.
Time Frame: Baseline and at the end of each 21-day Cycle assessed up to 32 months (final study analysis)
Population: The analysis population includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vorinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 317 | 320
Months | 7.73 (7.00) [7.00 to 8.53] | 7.03 (6.33) [6.33 to 7.73]

5. Secondary Outcome: Objective Response Rate
Description: Objective response rate was measured as the proportion of patients who achieved a confirmed partial response or better during the course of the study. Response to study therapy was assessed using EBMT Criteria and confirmed by Independent Adjudication Review.
Time Frame: Baseline and at the end of each 21-day Cycle assessed up to 32 months (final study analysis)
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vorinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 315 | 320
Percentage of Participants | 56.2 (50.5) [50.5 to 61.7] | 40.6 (35.2) [35.2 to 46.2]

ADVERSE EVENTS:
Time Frame: Up to 722 days.
Description: Adverse events were reported for the All Participants as Treated Population that included all randomized participants who received at least one dose of study treatment.
Arm/Group | Vorinostat + Bortezomib | Placebo + Bortezomib
Serious Adverse Events (participants affected / at risk) | 130/315 | 138/320
Other Adverse Events (participants affected / at risk) | 312/315 | 306/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat + Bortezomib (N=315) | Placebo + Bortezomib (N=320)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (13) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (3)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 9 (12) | 10 (10)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (8) | 7 (8)
Asthenia (General disorders) | 2 (2) | 1 (1)
Death (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 3 (3) | 5 (6)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pelvic mass (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (7) | 9 (12)
Swelling (General disorders) | 1 (1) | 0 (0)
Hepatic necrosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3)
Bronchitis pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 4 (4) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (3) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 6 (9) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 6 (6)
Herpes zoster ophthalmic (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 14 (17) | 13 (13)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 3 (4)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 32 (52) | 27 (43)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 13 (13)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic coma (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 4 (4)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 4 (5)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat + Bortezomib (N=315) | Placebo + Bortezomib (N=320)
Anaemia (Blood and lymphatic system disorders) | 91 (198) | 79 (164)
Leukopenia (Blood and lymphatic system disorders) | 42 (121) | 32 (122)
Neutropenia (Blood and lymphatic system disorders) | 112 (406) | 95 (300)
Thrombocytopenia (Blood and lymphatic system disorders) | 172 (749) | 106 (384)
Abdominal distension (Gastrointestinal disorders) | 8 (11) | 17 (21)
Abdominal pain (Gastrointestinal disorders) | 22 (37) | 27 (40)
Abdominal pain upper (Gastrointestinal disorders) | 26 (42) | 13 (20)
Constipation (Gastrointestinal disorders) | 64 (91) | 86 (132)
Diarrhoea (Gastrointestinal disorders) | 194 (604) | 133 (275)
Dyspepsia (Gastrointestinal disorders) | 24 (38) | 26 (40)
Nausea (Gastrointestinal disorders) | 193 (457) | 126 (247)
Vomiting (Gastrointestinal disorders) | 140 (280) | 80 (127)
Asthenia (General disorders) | 46 (89) | 40 (80)
Fatigue (General disorders) | 125 (350) | 96 (176)
Oedema peripheral (General disorders) | 24 (28) | 24 (27)
Pyrexia (General disorders) | 66 (114) | 70 (130)
Herpes zoster (Infections and infestations) | 22 (26) | 19 (21)
Nasopharyngitis (Infections and infestations) | 16 (22) | 18 (20)
Upper respiratory tract infection (Infections and infestations) | 55 (76) | 38 (58)
Blood creatinine increased (Investigations) | 17 (26) | 11 (14)
Weight decreased (Investigations) | 22 (36) | 22 (30)
Decreased appetite (Metabolism and nutrition disorders) | 75 (123) | 85 (139)
Hypokalaemia (Metabolism and nutrition disorders) | 35 (57) | 25 (40)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (34) | 27 (40)
Back pain (Musculoskeletal and connective tissue disorders) | 49 (67) | 47 (69)
Bone pain (Musculoskeletal and connective tissue disorders) | 15 (27) | 24 (39)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 (25) | 15 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (21) | 38 (52)
Dizziness (Nervous system disorders) | 36 (56) | 27 (37)
Dysgeusia (Nervous system disorders) | 23 (28) | 6 (8)
Headache (Nervous system disorders) | 35 (45) | 34 (45)
Hypoaesthesia (Nervous system disorders) | 10 (12) | 18 (26)
Neuralgia (Nervous system disorders) | 82 (124) | 86 (125)
Neuropathy peripheral (Nervous system disorders) | 62 (94) | 64 (97)
Paraesthesia (Nervous system disorders) | 20 (27) | 12 (14)
Peripheral sensory neuropathy (Nervous system disorders) | 33 (58) | 27 (39)
Insomnia (Psychiatric disorders) | 28 (32) | 29 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 52 (71) | 48 (61)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 (36) | 28 (35)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 13 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 24 (26) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 31 (43) | 40 (61)
Hypertension (Vascular disorders) | 29 (37) | 13 (16)
Hypotension (Vascular disorders) | 19 (23) | 12 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An investigator may not independently publish the results for their study site until after the multicenter publication, or 24 months after completion of study.

Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.